CLINICAL TRIAL: NCT06702176
Title: "Using a Multisite TENS System (Transcutaneous Electrical Noninvasive Stimulation) to Improve Fibromyalgia-related Symptoms (EXOFIB 3)"
Brief Title: "Using a Multisite TENS SysteM to Improve Fibromyalgia-related Symptoms.
Acronym: EXOFIB3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut De La Colonne Vertebrale Et Des Neurosciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-A00019-38
Record Dates: First submitted 2024-11-02; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-03

CONDITIONS: Fibromyalgia, Pain
Keywords: Exopulse Mollii Suit, Fibromyalgia
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Intervention Model Description: The investigators designed a trial that includes two phases: (i) phase 1 which consists of a 2-week intervention of Exopulse Mollii suit "active" versus "sham", separated by a 2-week washout period to prevent any carry-over effects; (ii) phase 2 that will be carried out two weeks following the end of phase 1. Phase 2 will last 6 months (24 weeks: 7 sessions per week) with a monthly assessment aiming to explore the long-term effects of this method on fibromyalgia.
  Summary:
  * Phase 1: randomized sham-controlled crossover study (active vs. sham condition/ assessment every two weeks )
  * Phase 2: Open-label (active condition, 6 months/monthly assessment)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Condition (Active Comparator): Active sessions will last 1 hour each. The following parameters will be used for electric stimulation: low frequency (20 Hz), low current intensity (2 mA), with a small pulse width of 25-170 microseconds. These parameters were previously found to be safe in human studies.
  Interventions: Device: EXOPULSE MOLLII SUIT active
- Control Condition (Sham Comparator): The control arm will be a sham intervention. The patients will receive a sham stimulation, for which the same Exopulse Mollii suit will be used but the control unit will be programmed to start stimulating for 1 minute then it will shut off which could enable cutaneous sensations that mimic the active condition, aiming to achieve an effective blinding integrity. There is no risk related to the sham intervention since it consists of applying the same parameters used for the active session (low frequency: 20 Hz; current intensity: 2 mA; pulse width ranging from 25 to 170 µs) but for a shorter duration of time (1 minute).
  Interventions: Device: EXOPULSE MOLLII SUIT (sham)

INTERVENTIONS:
Device: EXOPULSE MOLLII SUIT active — Exopulse Mollii suit is a new assistive device that has been developed by Exoneural Network (initially Inerventions AB), a Swedish med-tech company. Exopulse Mollii suit is a full-body garment with integrated 58 electrodes that can transcutaneously stimulate several groups of muscles. The device is CE labelled and is intended to use for reducing spasticity and improving blood circulation. The outfit is very easy to put on, it can be used for one hour every day and the analgesic effects last 24 hours or more. EXOPULSE Mollii suit consists of transcutaneous stimulation of several muscles by means of a feeble electric current (i.e., low frequency ~20 Hz, low-intensity 2mA), aiming to reduce pain. This treatment method theoretical background primarily refers to the theory of gate control. Based on this theory, the stimulation of large proprioceptive fibers would inhibit the nociceptive information transmitted by small fibers.
  Arms: Experimental Condition
Device: EXOPULSE MOLLII SUIT (sham) — It consists of applying the same parameters used for the active session (low frequency: 20 Hz; current intensity: 2 mA; pulse width ranging from 25 to 175 µs) but for a shorter duration of time (1 minute).
  Arms: Control Condition

SUMMARY:
Fibromyalgia is a debilitating pain condition that is characterized by the chronic occurrence of pain affecting the musculoskeletal system, a sensitivity to pressure stimuli, and a low threshold to noxious stimuli. The topography of pain is widespread, although it could be more pronounced in some bodily regions. Besides pain, patients suffer from a wide range of symptoms, including fatigue, anxiety and depression manifestations, and altered quality of life. Facing these debilitating symptoms, the available therapeutic strategies for treating pain and associated manifestations are usually faced with limited efficacy and numerous side effects. A previous pilot trial on fibromyalgia (EXOFIB-1 study) was conducted to evaluate the effects of Exopulse Mollii suit on fibromyalgia has showed beneficial and promising results. The intervention significantly alleviated pain, reduced fatigue, decreased physical and psychosocial impact of the disease, and improved the quality of life of patients with fibromyalgia. However, the observed effect sizes were small to medium. The investigators believe that a stimulation duration extended to six months would yield more positive outcomes and higher effect magnitude.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 75 years, with a definite diagnosis of fibromyalgia according to the American College of Rheumatology (ACR) 2010 criteria, set for at least three months
* Patients should be French speakers, able to understand verbal instructions, and affiliated with the National Health insurance

Exclusion Criteria:

* Patient included in another research protocol during the study period
* Patient unable to undergo medical monitoring for the study purposes due to geographical or social reasons
* Patient with contraindication to wearing Exopulse Mollii suit (e.g., cardiac stimulator, a ventriculoperitoneal shunt, intrathecal baclofen pump, pregnancy, and/or body mass index above 35 kg/m2)
* Patient with somatic or psychiatric diagnoses other than anxiety and depression (e.g., arrhythmias, uncontrolled epilepsy, other diseases causing osteoarticular and muscular pain)
* Any change in the pharmacological therapy in the last three months
* Introduction of a medical device other than Exopulse Mollii suit during the study period
* Patient under juridical protection (" mesure de protection judiciare : tutelle, curatelle, sauvegarde de justice ")

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Reduction of functional disability as per the Fibromyalgia Impact Questionnaire (FIQ) right after the intervention (phase 1) | This will be assessed before and after each condition (phase 1, 1 session per condition sham or active stimulation) at Visit 1(Day 0) ,Visit 2 (Day 15), Visit 3( Day 30) and Visit4 (Day 45)
  It is an 11-item scale that provides the researchers with a global assessment of the fibromyalgia syndrome, by measuring assesses Quality of Life and measures health status and functional disability and by exploring the impact of fibromyalgia on work, wellbeing, fatigue, sleep, stiffness, anxiety, and depression. FIQ ( Fibromyalgia Impact Questionnaire) scores can range from 0 to 100, with higher scores reflecting worse health status. Scores could be used to classify fibromyalgia as mild (scores: 0- 38), moderate (scores: 39-58), and severe (scores: 59-100)

SECONDARY OUTCOMES:
Reduction of functional disability as per the Fibromyalgia Impact Questionnaire (FIQ) throughout the follow-up period (phase 2) | This will be assessed during the phase 2 visits (6 months of using the EXOPULSE Mollii suit). The visits will take place monthly, starting from visit 5 and throughout visits 6, 7, 8, 9, 10 and 11.
  The Fibromyalgia Impact Questionnaire (FIQ) is a brief 10-item, self-administered instrument that measures physical functioning, work status, depression, anxiety, sleep, pain, stiffness, fatigue, and well being.
Analgesic effects based on the Visual Analogue Scale (VAS) during phases 1 and 2. | This will be assessed through study completion, an average of 8 months (at Visits 1, 2, 3, 4, 5, 6,7,8,9,10 and 11).
  VAS (Visual Analogue Scale ) which consists of rating the symptom on a 10 cm horizontal line going from "no pain" to "worst pain imaginable".
  Moreover, patients will be asked to fill in a pain diary (average daily pain reporting using a VAS filled in at the end of the day) and a pain medication that will be used to track pain medication use (opioids and nonopioids) one week prior, during, and till two weeks after each block.
Analgesic effects based on the Brief Pain Inventory (BPI) during phases 1 and 2. | This will be assessed through study completion, an average of 8 months (at Visits 1, 2, 3, 4, 5, 6,7,8,9,10 and 11).
  The validated French version of the Brief Pain Inventory (BPI) will be used to assess pain severity (4 items) and pain interference (7 items).BPI items are rated on a 10-point scale running from 0 (no pain/does not interfere) to 10 (pain as bad as possible/interferes completely).
Analgesic effects based on the Pain Catastrophizing Scale (PCS) during phases 1 and 2. | This will be assessed through study completion, an average of 8 months (at Visits 1, 2, 3, 4, 5, 6,7,8,9,10 and 11).
  The Pain Catastrophizing Scale (PCS) will also be employed, it is a valid and reliable scale that includes 13 items assessing the presence and severity of feelings or thoughts that emerge when experiencing pain. Each item is rated on a 5-point Likert scale ranging from 0 (not at all) to 4 (all the time).
Anti-fatigue effects according to the Visual Analogue Scale (VAS Fatigue) during phases 1 and 2. | This will be assessed through study completion, an average of 8 months (at Visits 1, 2, 3, 4, 5, 6,7,8,9,10 and 11).
  Like pain, fatigue will be assessed using VAS fatigue (Visual Analogue Scale)
Mood changes as per the Hospital Anxiety and Depression Scale (HADS) (phases 1 and 2) | This will be assessed through study completion, an average of 8 months (at Visits 1, 2, 3, 4, 5, 6,7,8,9,10 and 11).
  It is a 14-item generic scale with good psychometric properties. It consists of seven items assessing anxiety and seven others assessing depression. Scores can range from 0 to 21 on each subscale, with higher scores indicating worse symptomatology.
Quality of life using the Short Form 36 Health Survey (SF-36) during phases 1 and 2 | This will be assessed through study completion, an average of 8 months (at Visits 1, 2, 3, 4, 5, 6,7,8,9,10 and 11).
  It is a generic survey that contains 36 items that assess the quality of life and yield eight dimensions: physical functioning, physical role, emotional role, bodily pain, general health, vitality, social functioning, and mental health. The score of each dimension ranges from 0 to 100, with higher scales implying better health status.
Sleep changes using the Leeds Sleep Evaluation Questionnaire (LSEQ) during phases 1 and 2. | This will be assessed through study completion, an average of 8 months (at Visits 1, 2, 3, 4, 5, 6,7,8,9,10 and 11).
  Leeds Sleep Evaluation Questionnaire (LSEQ): it consists of 10 items that evaluate four domains: ease of initiating sleep, quality of sleep, ease of waking, and behavior following wakefulness. It is an easy-to-implement questionnaire that has been widely used to evaluate the subjective aspect of sleep. It has been employed in a large amount of psychological and psychopharmacological studies.
Sleep changes using the Pittsburgh Sleep Quality Index (PSQI) during phases 1 and 2. | This will be assessed through study completion, an average of 8 months (at Visits 1, 2, 3, 4, 5, 6,7,8,9,10 and 11).
  The Pittsburgh Sleep Quality Index (PSQI): it is a self-rated questionnaire that evaluates sleep quality. Its 19 questions aim to assess the sleep pattern during the previous month. This scale has good psychometric properties and its utility in clinical practice and research activities has been proven.
Evaluation of overall improvement using the CGI (Clinical Global Impression) | This will be assessed at visit 2 (day 15), visit 4 (day 45), and monthly from the second phase of 6 months of treatment (V5, V6, V7, V8, V9, V10, and V11), as the CGI is designed to be applied after the interventions.
  It consists of 7-point scale ranging from "very much improved since the initiation of treatment" to "very much worse since the initiation of treatment" (from 1 to 7)
Evaluation of patient's blinding to the type of stimulation in the crossover trial | This will only be assessed at Visit2 (Day 15) and Visit4 (Day 45) of Phase 1.
  This blind evaluation will be done in phase 1 using a dedicated questionnaire (only for each treatment condition, since all patients will receive the same active treatment in open phase 2).

CONTACTS AND LOCATIONS:
Overall Officials: Samar S Ayache, MD, PhD, HDR, Principal Investigator — Hopital Henri Mondor, Assistance Publique - Hôpitaux de Paris, Créteil, France
Locations (1):
- linical Neurophysiology department, Henri Mondor Hospital, Créteil, France, Créteil, VAL DE MARNE, France